CLINICAL TRIAL: NCT01748071
Title: Study of Analgesic Effect and Individual Sensitivity Differences of Opioid Analgesics
Brief Title: The Realtime Detection for Individual Variation of Analgesic ：A Comparison of Sufentanil vs Fentanyl
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang, Professor, MD., Huazhong University of Science and Technology
Other Study IDs: Individual Variation
Record Dates: First submitted 2012-12-09; First posted 2012-12-12 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: Surgery; Individuality
Keywords: fentanyl; sufentanil; individual variation; pain threshold; nacro-trend index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Sufentanil group: Grouped by intravenous injection of sufentanil at the time of anesthesia induction
- Fentanyl group: Grouped by intravenous injection of fentanyl at the time of anesthesia induction
- Saline group: Grouped by intravenous injection of saline before the time of anesthesia induction

SUMMARY:
Purpose: This study aimed to find a quick and timely way to investigate the individual variation of efficacy of opioid analgesic in Chinese patients undergoing elective surgeries. Methods: 120 female patients receiving elective surgery under general anesthesia were recruited into this study. At the time of routine intravenous anesthetic induction we observe the efficacy of opioid analgesic including analgesic effect, effects on Narco-trend index, sedative effect, effects on respiratory system, and aslo effects on cardiovascular system.

DETAILED DESCRIPTION:
Patients with the following diseases were excluded: known history of chronic pain, psychiatric diseases or communication disorders, diabetes mellitus, severe cardiovascular diseases, kidney or liver diseases with poor hepatic function, alcohol or drug abuse, heavy smoker, pregnancy or at the lactation period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65 years
* Anesthesiologists (ASA) physical status I or II;
* Within ±20% of ideal body weight;
* Agreed to participate the research

Exclusion Criteria:

* History of chronic pain;
* Psychiatric diseases;
* Diabetes mellitus;
* Severe cardiovascular diseases;
* Kidney or liver diseases;
* Alcohol or drug abuse (according to the criteria of DSM-IV);
* Pregnancy or at lactation period;
* Disagree to participate to the research

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 Chinese female patients receiving elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xianwei, MD, Study Director — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group
Started | 40 | 40 | 40
Completed | 38 | 38 | 40
Not Completed | 2 | 2 | 0
Not completed — Adverse Event | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 40 | 120
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (12) | 47 (13) | 49 (11) | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 40 | 120
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Mean Pressure Pain Threshold
Description: According to the measurement of pressure pain threshold after intravenous injection of opioid analgesics
Time Frame: 10 minutes after the procedure
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group
Number analyzed (Participants) | 38 | 38 | 40
kg/cm2 | 9.93 (3.50) | 6.20 (3.00) | 2.36 (0.97)

2. Primary Outcome: Mean Value of Narco-trend Index
Description: According to the measurement of Nacro-trend index after intravenous injection of opioid analgesics. Narco-trend index is from 0 to 100 which 0 represent deep sedation, and 100 represent waking state.
Time Frame: 10 minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group
Number analyzed (Participants) | 38 | 38 | 40
units on a scale | 50.9 (18.3) | 70.4 (27.3) | 93.7 (11.8)

3. Secondary Outcome: Mean Arterial Pressure
Description: According to the measurement of mean arterial pressure before and after intravenous injection of opioid analgesics
Time Frame: 10 minutes after the procedure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group
Number analyzed (Participants) | 38 | 38 | 40
mmHg | 90.1 (9.7) | 89.7 (12.8) | 90.3 (14.0)

4. Secondary Outcome: Mean Heart Rate
Description: According to the measurement of heart rate before and after intravenous injection of opioid analgesics
Time Frame: 10 minutes after the procedure
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group
Number analyzed (Participants) | 38 | 38 | 40
beats per minute | 77.9 (10.1) | 74.4 (12.9) | 77.6 (13.9)

5. Secondary Outcome: Mean Respiratory Frequency
Description: According to the measurement of respiratory frequency after intravenous injection of opioid analgesics
Time Frame: 10 minutes after the procedure
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group
Number analyzed (Participants) | 38 | 38 | 40
breaths per minute | 13.9 (3.3) | 12.3 (2.2) | 16.1 (3.1)

ADVERSE EVENTS:
Arm/Group | Sufentanil Group | Fentanyl Group | Saline Group
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/40

LIMITATIONS AND CAVEATS:
Because 3 patients couldn't maintain the SPO2 at 90% and 1 patient was at deep sedation, 4 subject patients were not analysed in the final results. These patients were performed as a routine intravenous anesthetic induction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes